CLINICAL TRIAL: NCT00729612
Title: Phase II Trial of Abraxane Plus Carboplatin for Advanced NSCLC for Patients at Risk of Bleeding From VEGF Directed Therapies
Brief Title: Paclitaxel Albumin-Stabilized Nanoparticle Formulation and Carboplatin in Treating Patients With Stage IIIB, Stage IV, or Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Greg Otterson (Other)
Collaborators: National Comprehensive Cancer Network (Network); Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Greg Otterson, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-08059; NCI-2011-03196 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2008-08-06; First posted 2008-08-07 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Taxes; Immunoenzyme Techniques; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (nab-paclitaxel, carboplatin) (Experimental): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes and carboplatin IV over 1-2 hours on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carboplatin; Drug: paclitaxel albumin-stabilized nanoparticle formulation; Genetic: protein expression analysis; Other: immunoenzyme technique; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel albumin-stabilized nanoparticle formulation
Genetic: protein expression analysis
Other: immunoenzyme technique
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well paclitaxel albumin-stabilized nanoparticle formulation given together with carboplatin works in treating patients with stage IIIB, stage IV, or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the response rate, in terms of overall response rate (complete response and partial response), of paclitaxel albumin-stabilized nanoparticle formulation and carboplatin in patients with stage IIIB-IV or recurrent non-small cell lung cancer who are ineligible for treatment with bevacizumab.

Secondary

* To evaluate safety of this regimen in these patients.
* To describe the overall survival of these patients.
* To describe progression-free survival of these patients.

Tertiary Objectives

* To explore, in a pilot fashion, the activity of this regimen using predictive biomarkers including serum SPARC levels, methylation of SPARC in primary tumor samples and serum, Ras mutations, ERCC1 and SPARC immunohistochemistry, and serum miRNA expression profiles.

OUTLINE: Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes and carboplatin IV over 1-2 hours on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Paraffin-embedded tissue blocks or unstained slides and blood samples are collected for correlative studies. Samples are analyzed for serum SPARC by ELISA, Ras mutations, ERCC1 AND SPARC by immunohistochemistry, and serum miRNA expression profiling.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced non-small cell lung cancer (NSCLC) meeting 1 of the following criteria:

  * Stage IIIB disease with malignant pleural effusion
  * Stage IV disease
  * Recurrent disease
* Squamous cell histology allowed
* Not eligible for curative treatment or treatment with bevacizumab
* Measurable disease according to RECIST
* Tumor (paraffin blocks or slides) must be available for correlative biomarker studies
* No uncontrolled brain metastases (or leptomeningeal disease)

  * Controlled brain metastases allowed

    * Able to receive appropriate therapeutic radiotherapy
    * Able to taper off all steroids without symptoms suggestive of increased intracranial pressure (nausea, vomiting, focal neurologic symptoms) for at least 7 days

PATIENT CHARACTERISTICS:

* ECOG (Eastern Cooperative Oncology Group) performance status 0-2
* ANC (absolute neutrophil count) ≥ 1.5 x 10^9/L
* Platelets ≥ 100 x 10^9/L
* Hemoglobin ≥ 9.0 g/L
* Total bilirubin ≤ 1.5 mg/dL
* AST (aspartate aminotransferase) and ALT (alanine aminotransferase) < 2.5 times upper limit of normal
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance > 50 mg/mL
* No known HIV or hepatitis B or C
* Not pregnant
* Negative pregnancy test
* Thrombotic or embolic event within the past 6 months allowed, provided adequately controlled with therapeutic anticoagulation
* Hemoptysis allowed, provided it is not life threatening or requires palliative procedures (e.g., endobronchial therapy or radiotherapy)
* No cardiac disease, including any of the following:

  * NYHA (New York Heart Association) class III-IV congestive heart failure
  * Unstable angina (angina symptoms at rest)
  * New onset angina (began within the past 3 months)
  * Myocardial infarction within the past 6 months
* No uncontrolled hypertension, defined as systolic blood pressure (BP) > 150 mm Hg or diastolic BP > 90 mm Hg despite optimal medical management
* No peripheral neuropathy ≥ grade 2
* No active clinically serious infection > CTCAE grade 2
* No serious non-healing wound, ulcer, or bone fracture
* No significant traumatic injury within the past 4 weeks
* No evidence or history of bleeding diathesis or coagulopathy
* No prior malignancy, except for adequately treated basal cell skin cancer, carcinoma in situ of the cervix, or other cancer for which the patient has been disease-free for 2 years

  * Stage I (T1c) prostate cancer adequately treated 2 years prior to diagnosis of NSCLC allowed, however metastatic prostate cancer currently receiving hormonal therapy or chemotherapy is not allowed
* No significant psychiatric illness, in the opinion of the principal investigator, that would prevent adequate informed consent or render therapy unsafe

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Concurrent therapeutic anticoagulation, > 325 mg acetylsalicylic acid, or chronic non-steroid anti-inflammatory drug use allowed
* At least 14 days since prior and no concurrent radiotherapy
* More than 4 weeks since prior major surgery or open biopsy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-08-14 (Actual); Primary Completion 2011-12-16 (Actual); Study Completion 2011-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A. Otterson, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Bertino EM, Williams TM, Nana-Sinkam SP, Shilo K, Chatterjee M, Mo X, Rahmani M, Phillips GS, Villalona-Calero MA, Otterson GA. Stromal Caveolin-1 Is Associated With Response and Survival in a Phase II Trial of nab-Paclitaxel With Carboplatin for Advanced NSCLC Patients. Clin Lung Cancer. 2015 Nov;16(6):466-74. doi: 10.1016/j.cllc.2015.05.004. Epub 2015 May 13. PMID 26123189
- [Derived] Owen DH, Williams TM, Bertino EM, Mo X, Webb A, Schweitzer C, Liu T, Roychowdhury S, Timmers CD, Otterson GA. Homologous recombination and DNA repair mutations in patients treated with carboplatin and nab-paclitaxel for metastatic non-small cell lung cancer. Lung Cancer. 2019 Aug;134:167-173. doi: 10.1016/j.lungcan.2019.06.017. Epub 2019 Jun 17. PMID 31319977
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled in the trial between September 2008 and December 2011.
Period: Overall Study
Arm/Group | Treatment (Nab-paclitaxel, Carboplatin)
Started | 63
Died Before Cycle 1 | 1
Received Cycle 1 | 62
Did Not Receive Cycle 2 | 7
Received Cycle 2 | 54
Died After Cycle 2 Before Response Eval | 1
Completed | 53
Not Completed | 10
Not completed — Non evaluable for response | 10

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Nab-paclitaxel, Carboplatin): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes and carboplatin IV over 1-2 hours on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  carboplatin
  paclitaxel albumin-stabilized nanoparticle formulation
  protein expression analysis
  immunoenzyme technique
  immunohistochemistry staining method
  laboratory biomarker analysis
Arm/Group | Treatment (Nab-paclitaxel, Carboplatin)
Number analyzed (Participants) | 63
Age, Continuous [Median (Full Range); unit: years] | 63.3 [36 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 42
Region of Enrollment [Number; unit: patients]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate Defined as Complete or Partial Response as Assessed by RECIST Version 1.0 Criteria.
Description: Response rate is overall response rate (CR+PR) as defined by RECIST criteriaPer Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Nab-paclitaxel, Carboplatin)
Number analyzed (Participants) | 54
percentage of patients
  Partial Response | 38.1 [26.1 to 51.2]
  Complete Response | 0 [0 to 0]

2. Secondary Outcome: Progression Free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Nab-paclitaxel, Carboplatin)
Number analyzed (Participants) | 63
months | 5.0 [4.3 to 6.4]

3. Secondary Outcome: Overall Survival
Description: Will be analyzed using a Kaplan-Meier methods.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Nab-paclitaxel, Carboplatin)
Number analyzed (Participants) | 63
months | 9.7 [8.4 to 13.2]

4. Secondary Outcome: Incidence and Intensity of Adverse Events Graded According to NCI CTCAE v. 3.0
Description: The incidence and intensity of adverse events graded according to NCI CTCAE v. 3.0 will be evaluated using descriptive statistics
Time Frame: Up to 5 years
Population: Grade 3 and 4
Measure: Number; unit: patients
Arm/Group | Treatment (Nab-paclitaxel, Carboplatin)
Number analyzed (Participants) | 63
patients
  Anemia | 7
  Neutropenia | 12
  Thrombocytopenia | 7
  Leukopenia/lymphopenia | 13
  Sensory neuropathy | 19
  Fatigue | 14

ADVERSE EVENTS:
Description: All toxicities were assessed using Common Terminology for Adverse Events (CTCAE) version 3.0
Arm/Group | Treatment (Nab-paclitaxel, Carboplatin)
Serious Adverse Events (participants affected / at risk) | 2/63
Other Adverse Events (participants affected / at risk) | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nab-paclitaxel, Carboplatin) (N=63)
Dehydration (Gastrointestinal disorders) | 1 (1)
Death NOS (General disorders) | 1 (1) — NOS=not otherwise specified
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nab-paclitaxel, Carboplatin) (N=63)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Neutropenia (Blood and lymphatic system disorders) | 13 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (7)
Leukopenia/Lymphopenia (Blood and lymphatic system disorders) | 13 (13)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Sensory Neuropathy (Nervous system disorders) | 19 (19)
Dehydration (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 14 (14)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes